CLINICAL TRIAL: NCT04113954
Title: Detecting Compartment Syndrome Pain in the Presence of Regional Anesthesia in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Kristin Schreiber, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019P002781
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Compartment Syndrome of Leg; Healthy
Keywords: Healthy volunteer; Regional anesthesia; Compartment Syndrome
MeSH Terms: conditions — Compartment Syndromes | interventions — Mepivacaine; Prilocaine

STUDY DESIGN:
Intervention Model Description: Our patients will be randomized to one of six arms.
Who Masked: Participant
Masking Description: Participant will be masked to the drug being provided in the nerve blocks (0.375% mepivacaine or 1.5% mepivacaine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Leg 1 ACB + low dose SNB-PF (Experimental): Right leg and 0.375% mepivacaine popliteal fossa-sciatic
  Interventions: Drug: Mepivacaine Injection
- Leg 1 ACB + high dose SNB-PF (Experimental): Right leg and 1.5% mepivacaine popliteal fossa-sciatic
  Interventions: Drug: Mepivacaine Injection
- Leg 2 ACB + low dose SNB-PF (Experimental): Left leg and 0.375% mepivacaine popliteal fossa-sciatic
  Interventions: Drug: Mepivacaine Injection
- Leg 2 ACB + high dose SNB-PF (Experimental): Left leg and 1.5% mepivacaine popliteal fossa-sciatic
  Interventions: Drug: Mepivacaine Injection
- Leg 1 ACB only (Experimental): Right leg and 1.5% mepivacaine ACB
  Interventions: Drug: Mepivacaine Injection
- Leg 2 ACB only (Experimental): Left leg and 1.5% mepivacaine ACB
  Interventions: Drug: Mepivacaine Injection

INTERVENTIONS:
Drug: Mepivacaine Injection — Injection of 0.375% mepivacaine in nerve block
  Other Names: Prilocaine
  Arms: Leg 1 ACB + high dose SNB-PF; Leg 1 ACB + low dose SNB-PF; Leg 2 ACB + high dose SNB-PF; Leg 2 ACB + low dose SNB-PF
Drug: Mepivacaine Injection — Injection of 1.5% mepivacaine in nerve block
  Other Names: Prilocaine

SUMMARY:
The goal of the study is to determine how different types of Regional Anesthesia (nerve blocks) can be helpful to patients with lower extremity trauma who develop compartment syndrome (an increased pressure in the fascial compartments) which can occur after injury to the leg.

This is a prospective, randomized study in healthy volunteers, who will undergo testing of the leg using a cuff inflation system, involving quantitative sensory testing (QST), questionnaire completion, with ultrasound scanning and nerve blocks in a supervised, monitored setting (BWH Clinical Investigation Center).

Specific Aims

1. Determine the effect of adductor canal-saphenous nerve block (ACB) and popliteal-fossa nerve block (SNB-PF) vs no block on pressure and ischemic pain in a model of compartment syndrome.

   1. Hypothesis: There will be minimal or no change in pressure pain threshold and tolerance and pain ratings with ACB alone
   2. Hypothesis: There will be an increase in pressure pain threshold and tolerance and decrease in pain ratings with ACB plus popliteal-fossa nerve block (SNB-PF), compared to no block
2. Determine the concentration dependence of SNB-PF effect on pressure and ischemic pain by comparing increasing doses of local anesthetic.

   1. Hypothesis: There will be a greater increase in pressure pain threshold and tolerance and great decrease in pain ratings with 1.5% mepivacaine than with 0.375% mepivacaine.

DETAILED DESCRIPTION:
Please complete the survey (copy and paste into new link). https://redcap.partners.org/redcap/surveys/?s=D4A4TN9TDL We will not contact you if the survey is incomplete.

Please contact us via email (ykchen@partners.org) about this study with subject line "Interested in participating in Compartment Syndrome Study"

Screening and Enrollment:

Healthy volunteers will be recruited, and all interested individuals will be invited to contact study staff to hear more about the study requirements and undergo a brief phone screen to determine eligibility. After their initial phone screen with study staff, interested subjects meeting eligibility requirements will be provided with an electronic copy of the consent form, perform a video consent, and schedule a study visit, to be conducted in the Clinical Investigation Center at Brigham and Women's Hospital. A 5 hour, 1 office visit is required.

All subjects will also undergo a survey-based COVID screen within 24 hours prior to the study.

Study day:

Immediately upon arrival for their study appointment, the physician investigator will go through the consent form in detail with each potential participant, and they will also be given a chance to read it thoroughly and have questions answered. Special care will be taken during the consent process to ensure subjects are fully competent and understand the nature of the questionnaires and testing procedures, including a brief demonstration of the devices and testing done. If agreeable to the study procedures after having questions answered, participants will provide informed consent. Each participant will be assigned a random ID number, and data will be collected, entered, and analyzed by ID number only. The subject's status as a patient will be unaffected by his/her decision to participate. If subject decides against participation at this point, they will be reimbursed for their time ($20).

Enrolled participants will complete basic deidentified demographic, clinical, psychosocial, and pain questionnaires. Brief validated questionnaires will include the PROMIS anxiety, depression, and sleep disturbance short forms, Pain Catastrophizing Scale (PCS), situational pain catastrophizing scale (sPCS), Brief Symptom Index, Fibromyalgianess scale, Brief Pain Inventory, Positive and Negative Affect Schedule, and pain coping strategies questionnaire.

After completing questionnaires, subjects will lie on a stretcher, with head of bed elevated to 30-45 degree angle according to comfort, with legs and feet exposed for testing.

QST testing Pressure pain threshold: Pressure algometry is the most commonly used test for static mechanical pressure sensation in the skin and in deep tissues. Pressure algometers deliver a firm and quantifiable pressure through a flat base applied to the skin. The electronic pressure algometer that we will use (Wagner Instruments) is a hand-held algometer utilizing a pressure-sensitive strain gauge, covered by a 0.5 cm2 circular probe. The probe is covered with a soft polypropylene disk, to avoid injury to the skin. The pressure applied through the probe is transduced, amplified, and converted to electrical reading on a digital display. The pressure will be slowly increased (1 lb/s) and the participant will be asked to note when they first feel pain and when they want the pressure to stop , which will be recorded as the pressure pain threshold and tolerance, respectively.120 This process will be repeated on the trapezius and the forearm, alternating between sides of the body with 20 seconds between measurements.

Pin Prick: This tests the detection and intensity of sharp type pain. In addition, it is often used as a modality to test temporal summation of pain with repeated stimuli. The conductor of the test will touch the participant on the finger with weighted mechanical probes in ascending order (64 mN, 128 mN, 256 mN, 512 mN), making sure to keep the probe perpendicular to the skin, and allowing the full weight to be resting on this point (i.e. the weight moves within the barrel), but without touching the barrel/cylinder itself to the skin. The participant will be instructed to rate the pain (0-10) of each stimulation. The conductor will make note of the lowest weight pin prick the participant indicated caused a 1-3 out of 10 pain. Then the conductor will perform the test of temporal summation to repeated punctate stimuli, which is considered an index of central pain-faciliatory processes. The pin prick weight that the participant noted was a 1-3 out of 10 pain is applied to the skin of the dorsal fingers at a frequency of 1Hz. Ten stimuli are applied, and the patient will be asked to rate the sensation of pain from the fifth, and tenth stimulus, as well as 15 seconds after the end of the stimulus train (PAS). The wind-up phenomenon occurs with progressive increase evoked pain with repeated stimulation and represents an index of central sensitization. Testing order will be performed on each hand, bilaterally, and on each foot.

Pressure Pain Threshold Assessment:

Pressure pain will be assessed through response to cuff pressure algometry (CPA). Tonic, deep-tissue, mechanical stimulation will be applied using a Hokanson rapid cuff inflator, which allows specific calibrated pressures to by administered and held for defined time periods. Using an adjustable cuff (similar to standard blood pressure cuff) wrapped around the leg, centered around the largest diameter of the gastrocnemius muscle, pressure will be increased by turning a manual dial at a rate of approximately 10-20 mmHg/second until the subject first feels pressure, and thereafter at approximately 5-10 mmHg/s, at which time subject will be asked to note when they first start feeling pain and then when they feel as though the pain is a 4, 6, 8 and 10 out of 10 VAS score (0 = no pain, 10 = worst pain), after which the cuff will be immediately deflated. Participants will be given a break. Cuff pressure at each of these points will be recorded 3 times for each leg to determine baseline pain thresholds.

Ischemic Pain Assessment:

The cuff will be re-inflated to the subject's average pressure previously determined to produce 4 out of 10 pain for that leg, and held for 5 minutes. A pulse oximeter will be placed on the big toe to monitor ischemia (pulse oximetry wave expected to disappear). Subjects will be asked for pain score at rest every 30 seconds, and pain score on passive stretch of gastrocnemius every 60 seconds. The participant will be reminded immediately before cuff inflation that they may ask for the pressure cuff to be deflated at any time, in which case this time will be recorded. Subjects will be asked to indicate the presence of tingling (paresthesias), and will rate pain at rest 30 and 60 seconds following cuff deflation (painful after sensations), as well as pain with passive stretch of gastrocnemius at 60 seconds after cuff deflation.

There will be a 1 minute break, then the cuff pressure will be inflated to a pressure corresponding to the next pain level as initially identified on the averaged baseline testing (ex: if pressure 4/10 was 100 mmHg and 6/10 was 150 mmHg, cuff pressure will first be held at 100 mmHg and held for 5 minutes, followed by a 1 minute break, and then reinflated at 150 mmHg and held for 5 minutes, followed by 1 minutes break, etc.). The above procedure will be repeated for cuff pressure at 6/10, 8/10, and 10/10. This will be done first on the "control leg" and then on the "block leg" prior to the nerve block placement. Subjects will be reminded that they may discontinue the cuff inflation at any point, and the time of cuff inflation recorded.

IV placement:

A 20 g IV will be placed prior to the start of any nerve block procedure. Site of IV placement will be cleaned with alcohol swab and initially anesthetized with 1% lidocaine administered through a small needle to allow greater comfort with IV placement.

Nerve Blocks:

Saphenous Nerve Block (ACB):

Subjects will lie supine with block leg slightly abducted. Standard monitors will be applied for vital monitoring (continuous pulse oximetry, EKG, blood pressure cuff every 5 minutes), and this monitoring continued until 20 minutes after block completion. Using sterile technique (cleaning of skin with chloroprep, sterile gloves, mask, sterile cap, sterile needle, sterile ultrasound probe cover and sterile gel), an ultrasound-guided approach will be used to identify the saphenous nerve and surrounding sonographic landmarks (sartorius muscle, vastus medialis, femoral artery, femoral vein, and adductor magnus). With a small needle, a small skin wheal of 1 cc of 1% lidocaine will be used to anesthetize the skin. Afterwards a standard 21 g, 10 cm block needle will be inserted and directed under ultrasound guidance to the saphenous nerve location. Aspiration on block syringe will be performed to confirm that needle tip is not within a vascular structure to avoid intraarterial or venous injection of local anesthetic. Incremental injection (5 cc at a time) of 1.5% mepivacaine will follow, with a total of 10 cc (150 mg) deposited around the saphenous nerve.

Popliteal sciatic Nerve Block (SNB-PF): (for dual nerve block group only) Participant will lie supine, with leg elevated to allow access to posterior leg for US scanning. Using sterile technique, an ultrasound-guided approach will be used to identify the common peroneal nerve and tibial nerve at the level of the popliteal fossa, and surrounding sonographic landmarks (femur, popliteal artery, and popliteal vein). The common peroneal and tibial nerves will be followed proximally by scanning proximally along the leg with the ultrasound until they form a unitary nerve (sciatic). With a small needle, a small skin wheal of 1 cc of 1% lidocaine will be used to anesthetize the skin of the lateral level at this level. Afterwards a standard 21 g, 10 cm block needle will be inserted and directed under ultrasound guidance to the sciatic nerve. Aspiration on block syringe will be performed to confirm that needle tip is not within a vascular structure to avoid intraarterial or venous injection of local anesthetic. Incremental injection (5 cc at a time) of 0.375% or 1.5% mepivacaine will follow, with a total of 15 cc (56.25 mg or 225 mg) deposited around the sciatic nerve.

Expected timeline Pressure pain threshold assessment will take approximately 3 minutes and Ischemic pain assessment approximately 30 minutes (5 minutes per inflation pressure with 1 minute for rest in between). Each assessment will be taken at baseline and 20 minutes after nerve block completion to allow full effect. Ultrasound measures of compartment pressures will be assessed before, during, and after pressure and ischemic pain assessment.

Resolution of Nerve block: Nerve blocks with mepivacaine are expected to be resolved within 4-6 hours, but monitoring will continue beyond this time as some normal variation in resolution may occur between individuals. Subjects will only be given assistance with getting off stretcher/chair if needed for 4 hours after nerve block placement. Strength testing of target nerve groups in lower extremity will be confirmed before subject is allowed to walk independently. Subjects gait and walking will be assessed and confirmed to be ambulating safely before discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 65 years old
2. BMI < 35
3. Able to speak and understand English
4. Willingness to undergo psychophysical testing
5. Willingness to have nerve block performed

Exclusion Criteria:

1. Ongoing acute or chronic pain in lower extremities
2. Diagnosis of neuropathy
3. Diagnosis of diabetes
4. History of chronic opioid use (having an opioid prescription > 30 days)
5. Loss of any limb
6. Currently pregnant
7. Any skin conditions or breakdown of skin affecting lower extremities
8. Current history of peripheral arterial disease
9. History of blood clot in any lower extremity
10. Current smoking/vaping of nicotine or illicit substances including marijuana

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Pressure-pain threshold and tolerance | 2 hours
  Pressure (mmHg) in cuff corresponding to pain score 4, 6, 8, and 10 out of 10 based on visual analog scale (VAS)
Ischemic pain threshold and tolerance | 2 hours
  Cuff inflation to predetermined pressure (mmHg) corresponding to pain score of 4, 6, 8, and 10 out of 10 based on pressure-pain threshold, and held for up to 5 minutes. Pain scores recorded every 30 seconds, pain scores every 1minute with passive stretch of the gastrocnemius.
Ultrasound measurement of pressure in compartment in leg | 1 hour
  Measurement of ultrasonographic qualities of compartments in the leg using both standard imaging as well shear wave elastography in response to varying external pressure of probe (0-22mmHg) using an external load sensor attached to the probe handle during pressure testing and block recovery, in the absence and presence of a thigh cuff set to 70 mmHg (non-painful pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schreiber, MD/PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YK, Lirk P, Flowers KM, Colebaugh CA, Wilson JM, Zeballos J, Von Keudell A, Barrett KE, Vlassakov K, Schreiber KL. Impact of varying degrees of peripheral nerve blockade on experimental pressure and ischemic pain: adductor canal and sciatic nerve blocks in a human model of compartment syndrome pain. Reg Anesth Pain Med. 2022 Jul 20:rapm-2022-103671. doi: 10.1136/rapm-2022-103671. Online ahead of print. PMID 35858717